CLINICAL TRIAL: NCT04754438
Title: Comparing the Efficacy of an Electronically Delivered Cognitive Behavioural Therapy Program to a Mental Health Coaching Program for Generalized Anxiety Disorder
Brief Title: Comparing the Efficacy of E-CBT to Mental Health Coaching for GAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Principal Investigator, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6032033
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Generalized Anxiety Disorder
Keywords: Mental Health; Psychotherapy; Electronic; Internet; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The randomized trial intervention will provide e-CBT for GAD through the Online Psychotherapy Tool (OPTT), a secure, cloud-based, digital mental health platform. Participants will be randomly assigned to either an e-CBT program tailored to GAD or a mental health coaching program over 12 weeks to address their anxiety symptoms. In the e-CBT group, participants will complete pre-designed modules and homework assignments while receiving personalized feedback and asynchronous interaction with a therapist through the platform. There will be 12 weekly sessions that include approximately 30 slides each along with interactive content, delivered through OPTT. In the mental health coaching group, participants will have weekly interaction with a therapist through the chat function in OPTT where the coach will check in on the participant and touch on a specific subject each week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- e-CBT (Experimental): 12 weekly sessions of approximately 30 slides and interactive content, delivered through OPTT. The e-CBT module content mirrors in-person standard CBT content, including different weekly topics, general information, skill overviews, and homework. Participants are instructed to go through the content and complete homework at the end of the session which helps them practice skills they learned through that session. Homework is submitted through OPTT and reviewed by the therapist assigned to the participant, who will provide personalized feedback within three days of submission. Therapists have access to pre-designed session-specific feedback templates to use as a basic structure to write their feedback. By doing so, the time needed to respond to each patient is reduced and therefore the number of patients each therapist can handle increases.
  Interventions: Behavioral: e-CBT
- Mental Health Coaching (Experimental): Weekly interactions with the therapist using general questions on the following topics:
  Week 1 (Mood) Week 2 (Sleep) Week 3 (Activity) Week 4 (Hobbies) Week 5 (Friendship) Week 6 (New Events) Week 7 (Job/Study) Week 8 (Diet/Food) Week 9 (Books/Movies/Shows) Week 10 (Phone/Apps/Games) Week 11 (Habits) Week 12 (Accomplishments)
  Interventions: Behavioral: Mental Health Coaching

INTERVENTIONS:
Behavioral: e-CBT — Electronically delivered cognitive behavioural therapy
  Arms: e-CBT
Behavioral: Mental Health Coaching — Electronically delivered mental health coaching
  Arms: Mental Health Coaching

SUMMARY:
This study will compare the efficacy of an electronically-delivered cognitive behavioural therapy (e-CBT) program versus a mental health coaching program to treat generalized anxiety disorder (GAD). This randomized trial intervention will provide the e-CBT and mental health coaching for GAD through a secure, online platform. Participants will be between the ages of 18 and 65 years with a confirmed diagnosis of GAD according to the Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5). Participants will either be offered an e-CBT program tailored to GAD or an online mental health coaching program over 12 weeks to address their anxiety symptoms. e-CBT participants will complete pre-designed modules and homework assignments while receiving personalized feedback and asynchronous interaction with a therapist through the platform. Participants in the coaching group will be contacted weekly through the online platform's chat feature. Therapists will ask the participants a series of pre-designed questions that revolve around a different theme each week to prompt conversation. Using clinically validated symptomology questionnaires, the efficacy of the e-CBT program will be compared to the coaching group. These questionnaires will be completed at baseline, week 6, week 12, and at a 6-month follow-up. Questionnaires include the State-Trait Anxiety Inventory (STAI), the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF), the Generalized Anxiety Disorder - 7 Item (GAD-7), and the Depression Anxiety Stress Scale - 42 Item (DASS-42).

DETAILED DESCRIPTION:
This randomized trial intervention will provide e-CBT for GAD through the Online Psychotherapy Tool (OPTT), a secure, cloud-based, digital mental health platform. Participants (age: 18-65 years) will be randomly assigned to either an e-CBT program tailored to GAD or a mental health coaching program over 12 weeks to address their anxiety symptoms. In the e-CBT group, participants will complete pre-designed modules and homework assignments while receiving personalized feedback and asynchronous interaction with a therapist through the platform. The content of the e-CBT modules is designed to mirror in-person standard CBT for GAD. There will be 12 weekly sessions that include approximately 30 slides each along with interactive content, delivered through OPTT. Using clinically validated symptomology questionnaires, the efficacy of the e-CBT program will be evaluated. In the mental health coaching group, participants will have weekly interaction with a therapist through the chat function in OPTT where the coach will check in on the participant and touch on a specific subject each week.

Participants (n = 110; 50 e-CBT participants, 50 coaching) aged 18-65 years will be recruited at Queen's University from outpatient psychiatry clinics at both Kingston Health Sciences Centre sites (Hotel Dieu Hospital and Kingston General Hospital). Additional recruitment will occur from Providence Care Hospital, family doctors, physicians, clinicians, and self-referrals in Kingston, Ontario, Canada. Once informed consent is provided, participants will be evaluated by a psychiatrist on the research team through secure video appointments to make or confirm a diagnosis of a generalized anxiety disorder (GAD) using the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).

During the informed consent process, it is explained to all participants that this program is not a crisis resource and that they will not have access to their therapist at all times. In the case of an emergency, participants are directed to the proper resources (e.g., emergency department, crisis lines, etc.) and this event will be reported to the principal investigator of the study.

Both e-CBT modules and in-person CBT sessions are designed to instill constructive and balanced coping strategies in participants. During the program, the focus will be on essential thinking and behavioural skills to help the patients become more engaged in day-to-day activities. The focus of the sessions is placed on the connection between thoughts, behaviours, emotions, physical reactions, and the environment. The goal is to change how patients evaluate negative beliefs and thought processes and their relationship with depression. Our goal is to adjust the negative thinking so that participants can think about and adapt to the things that are happening to them. This allows them to adjust the way they behave and think about their problems in a way that is not as negative and replaces those thoughts and behaviours with potentially more realistic and productive ones.

The e-CBT care plan consists of 12 weekly sessions of approximately 30 slides and interactive content, delivered through OPTT. The e-CBT module content mirrors in-person standard CBT content, including different weekly topics, general information, skill overviews, and homework. Participants are instructed to go through the content and complete homework at the end of the session which helps them practice skills they learned through that session. Homework is submitted through OPTT and reviewed by the therapist assigned to the participant, who will provide personalized feedback within three days of submission. Therapists have access to pre-designed session-specific feedback templates to use as a basic structure to write their feedback. By doing so, the time needed to respond to each patient is reduced and therefore the number of patients each therapist can handle increases. On average, developing this feedback takes a therapist 15-20 minutes per patient. In addition to the weekly feedback, participants have the option to message their therapist through the platform throughout the week regarding any questions or concerns they may have.

Participants in the coaching treatment program will have weekly interactions with a therapist through the chat feature in OPTT. The therapist will reach out weekly using the following structured question prompts to initiate interaction with their patient:

Week 1 - Mood: Tell me about yourself. How have you been feeling lately? How has the pandemic affected your mood? What differences have you noticed in your mood compared to the past? Week 2 - Sleep: How have you been? Tell me about your week. I want to ask about your sleep. How many hours do you get? Do you feel rested? Do you think you need to make any changes to your sleep hygiene? Week 3 - Activity: How was your week? How has your anxiety level been? What do you usually do to stay active during the days? Are there any indoor activities you can do at your place? Have you been using any online exercise programs? Week 4 - Hobbies: What did you do in the past week? Do you have any hobbies? How long have you been doing them? Have you found any new activities that you enjoy recently? Week 5 - Friendship: How was your week? How has the pandemic affected your relationship with your friends? Have you stayed in touch with your close friends during the pandemic? How often do you interact with your friends? Week 6 - New Events: How have you been? Have there been any new events in the past weeks? Are you planning to do anything new this week? Are you planning to do anything new this week? Are you expecting to hear any news from your family/friends? Week 7 - Job/Study: How have you been? Tell me about your week. How are you managing your day-to-day responsibilities (e.g., job, school, personal, etc.)? Week 8 - Diet/Food: How was your week? Let's talk about your eating habits. How does your anxiety affect your appetite? Are you satisfied with your diet? How often do you cook? Do you prefer home-made food or take-out? Week 9 - Books/Movies/Television: How was your week? Has your anxiety affected your concentration? Do you like reading books? What is the last book you read? Are there any books you would recommend to your friends? What shows do you enjoy watching? What are some shows you would recommend to your friends? Week 10 - Phone/Apps/Games: Tell me about your week. How many hours a day do you usually spend on your phone? What is your favourite app? Do you play any games? What kinds of games do you like to play (e.g., board games, cards, video games, etc.)? Week 11 - Habits: How have you been? How was your week? What do you think are some of your healthy habits? What are some habits you would like to change? Week 12 - Accomplishments: How was your week? How did you find this program? Were the weekly check-ins helpful? Overall, was this program helpful for you? Why or why not Are you interested in 12 weeks of online cognitive behavioural therapy? Why or why not?

All therapists are research assistants hired by the principal investigator. They all undergo training in psychotherapy and additional training from a psychiatrist on the research team before any interaction with participants. During this training, therapists complete feedback on practice homework, which is reviewed by a psychiatrist on the research team to ensure adequate quality of work. All therapists are supervised by the lead psychiatrist, who is an expert in the area of electronically delivered psychotherapy. Feedback is always reviewed by the lead psychiatrist, before submission to the participants.

Participants will only be identifiable by an anonymous identification number and any hard copies of consent forms will be stored securely in a locked filing cabinet and destroyed 5 years after study completion. Participant data will only be accessible by the care providers directly assigned to the participant and only anonymized data will be provided to the analysis team members. Participants will have the option to withdraw from the study at any point and request for their data to be removed from the analysis.

OPTT is Health Insurance Portability and Accountability Act (HIPAA), Personal Information Protection and Electronic Documents Act (PIPEDA), and Service Organization Control - 2 (SOC-2) compliant. Additionally, all servers and databases are hosted in Amazon Web Service (AWS) Canada cloud infrastructure which is managed by Medstack to assure all provincial and federal privacy and security regulations are met. OPTT does not collect any identifiable personal information or Internet Protocol (IP) addresses for privacy purposes. OPTT only collects anonymized metadata to improve its service quality and provide advanced analytics to the clinician team. OPTT encrypts all data, and no employee has direct access to participant data. All encrypted backups will be kept in the S3 storage that is dedicated to Queen's University.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 years of age at the start of the study
* Diagnosis of GAD according to DSM-5 by attending psychiatrist on research team
* Competence to consent to participate
* Ability to speak and read English
* Consistent and reliable access to the internet

Exclusion Criteria:

* Active psychosis
* Acute mania
* Severe alcohol or substance use disorder
* Active suicidal or homicidal ideation
* Receiving another form of psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in symptoms (State-Trait Anxiety Inventory) | Week 0, week 6, week 12, 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-4, 4 being the worst.
Change in symptoms (Generalized Anxiety Disorder - 7 Item) | Week 0, week 6, week 12, 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-3, 3 being the worst.
Change in symptoms (Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form) | Week 0, week 6, week 12, 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-5, 5 being the best.
Change in symptoms (Depression Anxiety Scale - 42 Item) | Week 0, week 6, week 12, 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-3, 3 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, MD, FRCPC, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Results will be shared through conference presentations, workshops, and journal publications.

REFERENCES:
- [Derived] Stephenson C, Kumar A, Malakouti N, Nikjoo N, Jagayat J, Gizzarelli T, Patel C, Gutierrez G, Shirazi A, Yang M, Omrani M, Alavi N. Comparing the Efficacy of an Electronically Delivered Cognitive Behavioral Therapy Program to a Mental Health Check-In Program for Generalized Anxiety Disorder: Protocol for a Randomized Trial. JMIR Res Protoc. 2023 Sep 20;12:e48899. doi: 10.2196/48899. PMID 37587552
- See also: Publication — https://journals-sagepub-com.proxy.queensu.ca/doi/full/10.1177/07067437241261933